CLINICAL TRIAL: NCT02375685
Title: A Safety Open-label Study of Gevokizumab in the Treatment of Patients With Chronic Non-infectious Uveitis Disease, an eXtension Study. The EYEGUARD-X Study
Brief Title: Long-term Safety of Gevokizumab in the Treatment of Patients With Chronic Non-infectious Uveitis (EYEGUARD-X)
Acronym: EYEGUARD-X
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL3-78989-019; 2013-004973-29 (EudraCT Number)
Record Dates: First submitted 2015-02-16; First posted 2015-03-03 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Chronic Uveitis
Keywords: Uveitis; Non-infectious Uveitis; Intermediate Uveitis; Posterior Uveitis; Behçet's disease uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Uveitis, Posterior | interventions — gevokizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gevokizumab (Experimental)
  Interventions: Biological: Gevokizumab

INTERVENTIONS:
Biological: Gevokizumab

SUMMARY:
The objective of this study is to evaluate long-term safety of gevokizumab in patient with chronic non-infectious uveitis who previously well tolerated the study drug and may benefit from longterm treatment with gevokizumab.

ELIGIBILITY:
Inclusion Criteria:

* either completed participation to one of the following: CL3-78989-002 open-label extension, or X052130/CL3-78989-005 double-masked period or open-label period, or X052131/CL3-78989-006 double-masked period or open-label period, or currently benefiting from gevokizumab compassionate use after participation in gevokizumab uveitis studies
* Male or female, age ≥18 (or legal age of majority in the country) at selection.
* For subject with reproductive potential, a willingness to use highly effective contraceptive measures

Exclusion Criteria:

* Meeting criteria for discontinuation of any of gevokizumab uveitis previous study.
* Infectious uveitis and masquerade syndrome
* History of severe allergic or anaphylactic reaction to study drug administration during previous study or to gevokizumab or any of its excipient.
* Currently active infectious disease.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety endpoints (adverse events, ...) | 108 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- Lions Eye Institute, Nedlands, Australia
- Medical Competence, Vienna, Austria
- CHU-Hôtel Dieu, Nantes, France
- Universitätsklinikum, Tübingen, Germany
- Interbalkan Medical Center, Thessaloniki, Greece
- Ospedale San Raffaele, Milan, Italy
- AIBILI, Coimbra, Portugal
- Severance Hospital, Seoul, South Korea
- ICOF ( Institut Clinic d'Oftalmologia ), Barcelona, Spain
- Chang Gung Memorial Hospital-Linkou, Taoyuan District, Taiwan
- Fattouma Bourguiba University hospital, Monastir, Tunisia
- Istanbul University, Istanbul, Turkey (Türkiye)
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Result] Tugal-Tutkun I, Pavesio C, De Cordoue A, Bernard-Poenaru O, Gul A. Use of Gevokizumab in Patients with Behcet's Disease Uveitis: An International, Randomized, Double-Masked, Placebo-Controlled Study and Open-Label Extension Study. Ocul Immunol Inflamm. 2018;26(7):1023-1033. doi: 10.1080/09273948.2017.1421233. Epub 2018 Jan 25. PMID 29370572
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov/condition/behcet-disease
- See also: U.S. FDA Resources — http://clinicaltrials.gov/ct2/info/fdalinks